CLINICAL TRIAL: NCT01898455
Title: IntraNasal Evaporative Cooling for the Symptomatic Relief of Migraine and Cluster Headache
Brief Title: Intranasal Cooling for Cluster Headache and Migraine
Acronym: COOLHEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumbria Partnership NHS Foundation Trust (Other)
Collaborators: BeneChill, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPFT001
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Migraine; Cluster Headache
Keywords: Migraine; Cluster headache; headache
MeSH Terms: conditions — Migraine Disorders; Cluster Headache; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intranasal Cooling (Experimental): RhinoChill Intranasal cooling, administered for 20 minutes. 10 treatment sessions per participant.
  Interventions: Device: RhinoChill intranasal cooling

INTERVENTIONS:
Device: RhinoChill intranasal cooling — The RhinoChill device will be used to locally cool the posterior nasopharynx, surrounding tissues and vasculature using a variable cooling flow rate based on patient comfort and tolerance, for a maximum of 20 minutes. Local anaesthetic spray will be administered to patients if the nasal catheters or cooling is poorly tolerated.
  Other Names: RhinoChill; Intranasal cooling; transnasal cooling

SUMMARY:
This study will be looking at the clinical efficacy of using a intranasal evaporative cooling device in providing relief of the symptoms of migraine and cluster headache. It will involve using a nasal catheter to spray a liquid coolant into the nasal cavity where it evaporates and removes heat from the tissue, thereby cooling the tissue and the blood vessels which supply blood to the brain. This cooling effect will cause the blood vessels to constrict and it is thought that this may provide symptomatic relief in both these forms of headache. 10 migraine patients and 5 cluster headache patients will be enrolled in the study and will receive 10 treatments each, for a maximum of 20 minutes at a time. They will be monitored during the treatment and for two hours afterwards to assess headache severity and side effects. There will be a further follow up 2 months after the last treatment to assess for longer term side effects from the treatment.

ELIGIBILITY:
Inclusion Criteria:

* >18 Years old.
* Meets criteria for NICE guidelines diagnosis of cluster headache or chronic migraine
* Has not responded satisfactorily to migraine prophylaxis or standard analgesia
* Capable of giving informed consent

Exclusion Criteria:

* < 18 years of age
* Subject has history of other severe co-morbid illness which would prevent full participation in the study
* Inability to insert the nasal cannulae
* Known temperature sensitive disorder such as reynauds, cryoglobulinaemia
* Known oxygen dependency to maintain SaO2 >95%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
• Reduction of pain score and overall symptoms from baseline in Migraine/cluster headache sufferers | 20 minutes
  When a participant presents with headache, baseline assessments will be performed for pain, nausea and other recognised symptoms of migraine/cluster headache. The Rhinochill device will be used to provide transnasal cooling for a period of 20 minutes then reassessment of pain and other symptoms will be undertaken.

SECONDARY OUTCOMES:
Tolerance to Rhinochill cooling during maximum 20 minutes treatment | 20 minutes
  Visual/analogue pain score and visual/analogue discomfort score
Adverse events noted throughout treatment phase and during follow up | 1 year
  • Any adverse events noted during the treatment or following treatment and during routine follow up will be recorded and analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Vanderpol, MD, Principal Investigator — Cumbria Partnership NHS Foundation Trust
Locations (1):
- Neurosciences department, Penrith Hospital, Cumbria Partnership NHS Foundation Trust, Penrith, Cumbria, United Kingdom

REFERENCES:
- [Derived] Vanderpol J, Bishop B, Matharu M, Glencorse M. Therapeutic effect of intranasal evaporative cooling in patients with migraine: a pilot study. J Headache Pain. 2015 Jan 26;16:5. doi: 10.1186/1129-2377-16-5. PMID 25623151